CLINICAL TRIAL: NCT00242060
Title: The Utility of Functional and Morphologic MRI in the Detection of Prostate Cancer for Patients With Elevated PSA and Prior Negative Biopsy
Brief Title: Functional and Morphologic MRI in the Detection of Prostate Cancer in Patients With Prior Negative Biopsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 02-0065-C
Record Dates: First submitted 2005-10-18; First posted 2005-10-19 (Estimated); Last update posted 2010-07-15 (Estimated); Status verified 2010-07

CONDITIONS: Elevated PSA; Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

INTERVENTIONS:
Procedure: MRI

SUMMARY:
Prostate specific antigen (PSA) and digital rectal exam (DRE) are used to screen for prostate cancer. Patients with abnormal DRE or elevated PSA undergo transrectal ultrasound guided biopsy (TRUS-Bx). There are some men who have a normal TRUS-Bx despite persistent elevated PSA and may harbor occult prostate cancer. The purpose of this study is to determine if MRI using an endorectal coil, and advanced MRI methods called H1 MR Spectroscopy (MRS) and Dynamic MR Perfusion Imaging (dMRI) can help identify and localize prostate cancer in these patients and direct repeat TRUS-Bx to the most suspicious location in the prostate gland. 100 men, currently under observation with elevated PSA but negative TRUS-Bx will be enrolled in the study.

DETAILED DESCRIPTION:
Prostate specific antigen (PSA) and digital rectal exam (DRE) are used to screen for prostate cancer. Patients with abnormal DRE or elevated PSA undergo transrectal ultrasound guided biopsy (TRUS-Bx). There are some men who have a normal TRUS-Bx despite persistent elevated PSA and may harbor occult prostate cancer. The purpose of this study is to determine if MRI using an endorectal coil, and advanced MRI methods called H1 MR Spectroscopy (MRS) and Dynamic MR Perfusion Imaging (dMRI) can help identify and localize prostate cancer in these patients and direct repeat TRUS-Bx to the most suspicious location in the prostate gland. 100 men, currently under observation with elevated PSA but negative TRUS-Bx will be enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

* prior ultrasound biopsy of prostate showing no cancer or only single microfocus of cancer

Exclusion Criteria:

* contraindication to contrast enhanced endorectal coil MRI

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-11; Primary Completion 2008-04 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Masoom Haider, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Princess Margaret Hospital, Toronto, Ontario, Canada